CLINICAL TRIAL: NCT04147884
Title: A Study to Evaluate the Feasibility and Safety of the Millipede Transcatheter Annuloplasty Ring System in Patients With Functional Mitral Regurgitation: (Millipede Feasibility Study)
Brief Title: A Feasibility Study of the Millipede Transcatheter Annuloplasty Ring System in Patients With Functional Mitral Regurgitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S2436
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation Functional; Mitral Valve Disease; Cardiovascular Diseases
Keywords: Functional Mitral Regurgitation; Mitral Repair
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Mitral Valve Repair (Experimental): All subjects will receive mitral valve repair using the Millipede System
  Interventions: Device: Millipede Transcatheter Annuloplasty Ring System (Millipede System)

INTERVENTIONS:
Device: Millipede Transcatheter Annuloplasty Ring System (Millipede System) — The Millipede Transcatheter Annuloplasty Ring System is a repair device used for treating mitral valve regurgitation (MR). The system consists of several components: a transcatheter annuloplasty ring (implant) which remains in the body and a delivery system and intracardiac echocardiography catheter (imaging device) used to deliver the implant to the mitral valve.

SUMMARY:
To evaluate the feasibility and safety of the Millipede Transcatheter Annuloplasty Ring System in subjects with functional mitral regurgitation

DETAILED DESCRIPTION:
The Millipede Feasibility Study is a prospective, open-label, single-arm study to assess the safety and feasibility/performance of the Millipede Transcatheter Annuloplasty Ring System in subjects with functional mitral regurgitation. The study will include subjects with functional mitral regurgitation classified as moderate to severe (3+) or severe (4+) that are symptomatic (NYHA Class II-IV) despite guideline directed medical therapy in whom the local hearth team determines that surgery is not an option for mitral valve repair. Clinical follow-up will be required in hospital, 30 days, 90 days, 6 months, 12 months, and then annually through 5 years post-procedure. Subjects who have any part of the Millipede Transcatheter Annuloplasty Ring System introduced into the body but who do not end up with an implant will be followed through 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
* Subject has moderate to severe (3+) or severe (4+) functional mitral regurgitation confirmed by echocardiography core lab
* Subject is symptomatic (NYHA Class II-IV) despite guideline directed medical therapy, including CRT if indicated
* The local site heart team concurs that mitral valve surgery will not be offered as a first-line treatment option
* Subject is a candidate for annuloplasty based on the criteria below as assessed by the investigative site (and confirmed by the Case Review Committee [CRC]):

Left Ventricular Ejection Fraction (LVEF) ≥ 25% Left Ventricular End Diastolic Diameter (LVEDD) ≤ 65 mm Coaptation distance (i.e. tenting height) < 10 mm Absence of posterior wall aneurysm

Exclusion Criteria:

* Subject has severe calcification of the mitral annulus or leaflets or other anatomic features that make the subject unsuitable for annuloplasty with the Millipede System in the judgment of the treating physician or subject does not have suitable mitral annular diameter (determined by CT) as per the Instructions for Use
* Transfemoral venous and transseptal access determined not to be feasible
* Subject is on the waiting list for a transplant or has had a prior heart transplant
* Subject has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 30 days prior to study enrollment
* Subject has had any percutaneous coronary, carotid, or other endovascular intervention within 30 days prior to study enrollment
* Subject has had carotid surgery within 30 days prior to study enrollment
* Subject has had any open coronary or vascular surgery (other than carotid surgery) within 3 months prior to study enrollment
* Subject has had a cardiac resynchronization therapy (CRT) device implantation within 3 months prior to study enrollment
* Subject has untreated clinically significant coronary artery disease requiring revascularization
* Any planned cardiac surgery within the next 12 months
* Need for emergent or urgent surgery for any reason
* Subject has severe aortic valve stenosis and/or aortic valve regurgitation
* Subject has physical evidence of right-sided congestive heart failure (CHF) with echocardiographic evidence of moderate or severe right ventricular dysfunction and/or severe tricuspid valve regurgitation
* Subject has the presence of prosthetic heart valve in any position
* Subject has renal insufficiency (eGFR <20mL/min) and is not on dialysis
* Subject has a life expectancy less than 12 months
* Subjects in whom trans-esophageal echocardiography-Doppler assessment is contraindicated or in which mitral regurgitation is not measurable by Transthoracic Echocardiography (TTE)
* Subject has a prior history of atrial septal defect (ASD) closure or patient foramen ovale (PFO) closure
* Subject has fixed pulmonary artery systolic pressure > 70 mmHG
* Subject has known hypersensitivity or contraindication to protocol required procedural or post procedural medication (e.g., anticoagulation therapy) or hypersensitivity to nickel or titanium
* Subject has known hypersensitivity to contrast that cannot be adequately premedicated
* Female subject who is breast feeding or is pregnant and planning to become pregnant within the study period
* Subject is participating in another investigational drug or device study that has not reached its primary endpoint or subject intends to participate in another investigational device clinical trial within 12 months after index procedure
* Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis
* Subject has oxygen-dependent chronic obstructive pulmonary disease
* Subject has documented severe liver disease
* Subject has Hgb <8 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3
* Subject has any evidence of intracardiac thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Technical Success Endpoint | Index procedure exit from the catheterization laboratory
  Technical Success (measured at exit from the catheterization laboratory) is defined per Mitral Valve Academic Research Consortium (MVARC ). All of the following must be present:
  Absence of procedural mortality; and Successful access, delivery and retrieval of the device delivery system; and Successful deployment and correct positioning of the first intended device; and Freedom from emergency surgery or reintervention related to the device or access procedure.
Primary Safety Endpoint | 30 days post index procedure
  The composite (aggregate) of the following implant-related and/or delivery-related serious adverse events (SAEs) at 30 days post index procedure (based on MVARC definitions and adjudicated by an independent clinical events committee). The unit of outcome measure is % (n/N):
  * Mortality: all-cause
  * Stroke: disabling and non-disabling; Bleeding: life-threatening based MVARC scale
  * Major access site vascular complications
  * Major cardiac structural complications due to access-related issues
  * Acute kidney injury (AKI; ≤7 days post index procedure): based on the Acute Kidney Injury Network (AKIN) --System Stage 3 (including renal replacement therapy) or Stage 2
  * Myocardial infarction (MI; periprocedural [≤48 hours] or spontaneous [>48 hours])
  * Coronary ischemia requiring percutaneous coronary intervention (PCI) or coronary artery bypass graft
  * Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gooley, MBBS, PhD, Principal Investigator — Monash Health; Nicolas Van Mieghem, MD, PhD, Principal Investigator — Erasmus Medical Center; Susheel K Kodali, MD, Principal Investigator — New York-Presbyterian/Columbia University Medical Center
Locations (4):
- United States (3):
  - Tucson Medical Center Healthcare, Tucson, Arizona
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
- Monash Health, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html)